CLINICAL TRIAL: NCT01425983
Title: Dietary Intervention of Stress-Induced Neurovegetative Disorders in Men and Women With a Specific Amino Acid Composition With Micronutrients
Brief Title: Dietary Intervention of Stress-Induced Neurovegetative Disorders With a Specific Amino Acid Composition (asn01)
Acronym: asn01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyberg Vital GmbH (Industry)
Responsible Party: Principal Investigator, Doris Meister, Doris Meister, Sponsor-Investigator, Kyberg Vital GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kyberg-02
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Nervous System Disorder; Imbalance of Constituents of Food Intake
Keywords: stress; lability and irritative disturbances; dietary supplement; amino acid composition; psychological neurological questionnaire (PNF)
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- amino acid composition (asn01) (Active Comparator): Dietary supplement: specific amino acid composition with micronutrients
  Interventions: Dietary Supplement: amino acid composition (asn01)
- Sugar powder (Placebo Comparator): Placebo contains no amino acids and no micronutrients and is identical in appearance and solution properties.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: amino acid composition (asn01) — Amino acid composition with micronutrients, once a day (in the evening, 2 hours after dinner) content of a sachet mixed with 200 ml water.
  Duration: 12 weeks
  Other Names: Brand name: aminoplus neurostress
  Arms: amino acid composition (asn01)
Other: Placebo — Placebo; once a day (in the evening, 2 hours after dinner) content of a sachet mixed with 200 ml water.
  Placebo contains no amino acids and micronutrients and is identical in appearance and solution properties.
  Duration: 12 weeks
  Arms: Sugar powder

SUMMARY:
Psychosocial stress leads to altered neuroendocrine functions, such as serotonergic dysfunction, as well as alterations of the autonomic nervous system and the hypothalamic-pituitary-adrenal (HPA) axis activity resulting in an imbalance between inhibitory and excitatory neurotransmitters. Clinical consequences include, inter alia, neurovegetative disorders, higher resting heart rate, hypertension, depressive symptoms, sleep disturbances, irregular body-weight changes, and insulin resistance. Poor dietary intake of the essential amino acid L-tryptophane as a precursor to 5-hydroxytryptamine (HT, serotonin) increases sensitivity to stress.

It is therefore the investigators hypothesis that daily oral administration of an amino acid mixture (dosage 3.8 g/day) with micronutrients specifically designed to decrease neurovegetative disorders will target these neuroendocrine and metabolic alterations in adults with psychosocial stress. The principal endpoints will be a decrease in points in the psychological-neurological questionnaire (PNF).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 Years
* Psychological-Neurological Questionnaire (PNF): 30 - 50 Points

Exclusion Criteria:

* Age: < 18 and > 65 Years
* Psychological neurological questionnaire (PNF): < 30 and > 50 Points
* Resting heart rate: < 70/min
* Supplementation with dietary supplements or drugs which contains amino acids, vitamins and other micronutrients
* Therapy with antipsychotic drugs such as tranquilizer, antidepressants
* acute and chronic diarrhea
* Psychological-neurological or psychiatric therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Psychological neurological questionnaire (PNF) | 12-week dietary intervention
  Pre-post intervention changes in total number of points PNF

SECONDARY OUTCOMES:
Psychological neurological questionnaire (PNF) | 12-week dietary intervention
  Pre-post improvement in total number of points from the psychological-neurological questionnaire (PNF) about 10 Points or more
Salivary cortisol concentration (30 minutes after waking in the morning) | 12-week dietary intervention
  Absolute difference between cortisol concentration at baseline and 12 weeks
Salivary cortisol concentration (in the evening between 8 and 10 pm, 2 hours after dinner) | 12-week dietary intervention
  Absolute difference between cortisol concentration at baseline and 12 weeks
Serotonin concentration in blood | 12-week dietary intervention
  Absolute difference between serotonin concentration at baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Metzner, Professor MD, Principal Investigator — Bonn Education Association for Dietetics r.A., Cologne, Germany
Locations (1):
- Cardiological Outpatient Practice Elke Parsi, MD, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Chaborski K, Bitterlich N, Alteheld B, Parsi E, Metzner C. Placebo-controlled dietary intervention of stress-induced neurovegetative disorders with a specific amino acid composition: a pilot-study. Nutr J. 2015 May 6;14:43. doi: 10.1186/s12937-015-0030-3. PMID 25943490